CLINICAL TRIAL: NCT07021755
Title: Comparison Of The Effects Of Intranasal And Oral Midazolam Premedication On Sedation And Separation From Parents For Pediatric Patients
Brief Title: Use Of Midazolam In Premedication Of Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SBU-ANESTHESİA-DMY-01
Record Dates: First submitted 2024-11-30; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Separation, Family; Separation Anxiety
Keywords: midazolam; premedication; children
MeSH Terms: conditions — Anxiety, Separation | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intranasal midazolam (Experimental): Twenty minutes before anesthesia induction, the first group were given 0.25 mg/kg intranasal midazolam and named Group N (n=30). Intranasal midazolam was administered by the parent with a 2 ml injector with the needle removed, with half the dose given into one nostril and the other half into the other nostril, while the patient was lying supine.
  Interventions: Other: midazolam
- oral midazolam (Experimental): The second group were given 0.5 mg/kg oral midazolam and called Group O (n=30). Patients given oral midazolam drank the calculated midazolam dose mixed with 5 ml pulp-free fruit juice.
  Interventions: Other: midazolam

INTERVENTIONS:
Other: midazolam

SUMMARY:
: The aim of the study is to compare the effect of intranasal and oral midazolam administered for premedication to children of preschool age on hemodynamic parameters, sedation and separation from parents.

DETAILED DESCRIPTION:
Patients meeting with anesthesiologists before surgery for assessment and administration of premedication is important in terms of reducing morbidity and mortality linked to surgery and anesthesia. A study reported that 75% of children experience anxiety before surgery. This anxiety and worry observed in the pediatric patient group may cause tachycardia, hypertension and tachypnea due to increased catecholamine levels in the body and may cause aggressive reactions that are difficult to control. Additionally, it may make control of postoperative pain more difficult .

Several drugs are used before anesthesia to resolve surgical anxiety in pediatric patients and facilitate problem-free transfer to the operating room.

Midazolam is a benzodiazepine group drug, commonly used for preoperative medication for a long time. Reasons for it being chosen for premedication are that it ensure sedation and anxiolysis, has rapid onset of effect, and is more amnesic than diazepam . Though there are many routes to administer the drug, IM and IV routes are painful and frightening for patients. The premedication administration route must be acceptable for the child and not be traumatic. As a result, generally oral and intranasal routes are chosen for sedation of pediatric patients.

The aim of this study was to compare the effects of intranasal and oral midazolam, administered for premedication to preschool children, on hemodynamic parameters, sedation level and separation from parents, and in terms of complications.

The study was planned as prospective, randomized and single-blind research. After receiving permission from the ethics committee of our hospital (Haseki Clinical Research Ethics Committee No: 28.05.2009/10), the study included a total of 60 children aged 2-6 years in ASA ( Physical Status Classification System) I-II group, with elective surgery planned under general anesthetic. . Patients were allocated to two equal groups with the closed envelope method (Group O, n=30, 0.5 mg/kg oral midazolam; Group N, n=30, 0.25 mg/kg intranasal midazolam). Midazolam was administered 20 minutes before the operation. Vital signs and sedation score levels were recorded every 5 minutes. At the end of the 20th minute, the separation from parents score was assessed and recorded. Assessments were completed by an anesthesiologist who did not know the method of administration for premedication.

ELIGIBILITY:
Inclusion Criteria: - Children 2-6 years old

* ASA I-II group
* with elective surgery planned under general anesthetic.

Exclusion Criteria:

* Patients allergic to midazolam
* rhinorrhea
* respiratory system dysfunction like nasal polyp
* neurological or psychiatric disorder

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2009-12-01 (Actual); Study Completion 2009-12-01 (Actual)

PRIMARY OUTCOMES:
sedation | five minute
  The level of sedation was monitored every 5 minutes with the Ramsey sedation scale. Sedation scores of 1 and 2 were inadequate, while sedation scores of 3 and 4 were accepted as satisfactory

SECONDARY OUTCOMES:
separation from parents | twenty minutes
  Twenty minutes later, separation from parents was assessed with a four-stage scale and recorded. For separation from parents, scores of 1 and 2 were satisfactory and scores of 3 and 4 were inadequate

CONTACTS AND LOCATIONS:
Overall Officials: Ecder Ozenc, Study Director — ozencecder@hotmail.com
Locations (1):
- Haseki training and research hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No